CLINICAL TRIAL: NCT03255551
Title: Blood Pressure Lowering Effects of Amosartan Regarding Proviso in Patients With Hypertension: Prospective, Multicenter, Observational Study
Brief Title: Blood Pressure Lowering Effects of Amosartan Regarding Proviso iN Patients With High Blood Pressure
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Other Study IDs: LEARN BP
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amosartan — amosartan is a combination of amlodipine, which is a calcium channel blocker (CCB), and rozatan, an angiotensin II receptor antagonist (ARB), and is an antihypertensive agent

SUMMARY:
Blood Pressure Lowering Effects of Amosartan Regarding Proviso in Patients with Hypertension

DETAILED DESCRIPTION:
After taking Amozatan (AMS, amlodipine / rozanthin combination) in patients with essential hypertension, the percentage of patients who reached the mean systolic target blood pressure was evaluated

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension whose blood pressure is not adequately controlled by amlodipine or rosartan monotherapy
* In patients with stage 2 hypertension (SBP 160-179 mmHg), patients requiring a combination therapy to reach the target blood pressure
* Patients who were changed to amosartan while using other hypertensive agents

Exclusion Criteria:

* Patients with hypersensitivity to dihydropyridine derivatives of amosartan
* Women who are pregnant or who may be pregnant and breastfeeding
* Patients with severe hepatic dysfunction
* Patients with severe aortic stenosis
* Patients at risk of shock
* Patients participating in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Estimated total number of patients: 3,150 Estimated number of centers: 37
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Patients with essential hypertension evaluated the mean blood pressure after taking amosartan. | 6 month
  Blood Pressure Lowering Effects of Amosartan Regarding Proviso in Patients with Hypertension

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SH, Ryu KH, Lee NH, Kang JH, Kim WS, Park SW, Lee HY, Kim JJ, Ahn YK, Suh SY. Efficacy of fixed-dose amlodipine and losartan combination compared with amlodipine monotherapy in stage 2 hypertension: a randomized, double blind, multicenter study. BMC Res Notes. 2011 Oct 28;4:461. doi: 10.1186/1756-0500-4-461. PMID 22035131
- [Background] Law MR, Wald NJ, Morris JK, Jordan RE. Value of low dose combination treatment with blood pressure lowering drugs: analysis of 354 randomised trials. BMJ. 2003 Jun 28;326(7404):1427. doi: 10.1136/bmj.326.7404.1427. PMID 12829555
- [Background] Choi SM, Seo MJ, Kang KK, Kim JH, Ahn BO, Yoo M. Beneficial effects of the combination of amlodipine and losartan for lowering blood pressure in spontaneously hypertensive rats. Arch Pharm Res. 2009 Mar;32(3):353-8. doi: 10.1007/s12272-009-1307-x. Epub 2009 Apr 23. PMID 19387578